CLINICAL TRIAL: NCT03738774
Title: Addressing Post-Intensive Care Syndrome Among Survivors of COVID (APICS-COVID)
Acronym: APICS
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, James C. Jackson, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: IRB181120
Record Dates: First submitted 2018-11-07; First posted 2018-11-13 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Post Intensive Care Syndrome
Keywords: Post intensive care syndrome
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will assess the relationship between early unmet needs after hospital discharge and subsequent clinical outcomes among survivors of acute respiratory failure. The investigators hypothesize that early unmet needs are associated with poor outcomes at three months.

DETAILED DESCRIPTION:
Despite the accumulation of data documenting the reality of extensive functional impairments following ICU stay, the specific treatment needs of individuals experiencing Post-Intensive Care Syndrome (PICS) are not well known largely because of a relative lack of knowledge about the specific unmet needs of patients at risk for PICS at the time of hospital discharge. These possible needs include oxygen prescriptions, equipment for noninvasive ventilation, durable medical equipment prescriptions, coordination with government assistance and community health programs, physical or occupational therapy in the home or at an outpatient clinic, medications restarted or discontinued as appropriate.

This study will enrol individuals who were diagnosed with acute respiratory failure during an ICU admission and were discharged from the ICU alive. Once enrolled, participants' medical records will be reviewed for demographic and medical information. Questionnaires will be used to assess the participant's status prior to ICU admittance, including comorbidities, medications, physical functioning, quality of life, alcohol/smoking/substance use, social support and healthcare utilization. While in the ICU, participants will receive usual clinical care in this observational study. Data on mechanical ventilation, arterial blood gas values, acute respiratory distress syndrome (ARDS) diagnosis, delirium, and medical status will be collected. Information regarding the patients' postdischarge needs including medical equipment, medication, home care services, dialysis, appointments, counselling and referral will also be collected by reviewing the discharge note. Follow-up evaluations by phone call will occur at 1-4 weeks, 3 and 6 months following the ICU discharge. At 1-4 weeks, the investigators will evaluate, via phone call whether the patient's post-discharge needs are met. At 3 months and 6 months phone calls, standardized surveys will be used to assess mortality status, readmission, healthcare utilization, functional outcomes, quality of life, mental health status, coping and social support and return to work.

ELIGIBILITY:
Inclusion Criteria:

1. Respiratory failure:

   * Mechanical Ventilation via endotracheal tube/tracheostomy ≥ 24hrs
   * continuous positive airway pressure (CPAP), bilevel positive airway pressure (BIPAP) ≥ 24 consecutive hrs (provided for acute respiratory failure not for Obstructive Sleep Apnea or other stable use)
   * High flow nasal cannula ≥ 24 consecutive hrs (FIO2 ≥ 0.5 and flow rate ≥ 30 L/min)
2. Expected to be discharged home alive
3. Within the pandemic expansion cohort, COVID-19 status (defined as a positive result on an appropriately validated molecular diagnostic assay for infection with SARS-CoV-2) will be used to guide enrollment

Exclusion Criteria:

* Lack of informed consent
* Patient in the ICU < 24hrs
* Mechanical ventilation at baseline
* Residing at a medical institution at the time of hospital admission
* Homelessness
* Primary residence not in USA
* Prisoner
* More than mild dementia (either known diagnosis of moderate or worse dementia or Informant Questionnaire on Cognitive Decline in the Elderly (IQ-CODE) > 3.6; screening performed on patient > 50 years old or with family reports of possible memory decline)
* Patient on hospice at or before time of enrollment
* Patients who, based solely on pre-existing medical problems (such as poorly controlled neoplasm or other end-stage disease, including Stage IV heart failure or severe burns), would not be expected to survive six months in the absence of the acute respiratory failure.
* Patient with neurological injury either receiving treatment for intracranial hypertension or who are not expected to return to consciousness.
* Unable to communicate by telephone in English or Spanish
* Patients mechanically ventilated solely for airway protection or obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the ICUs and/or hospital wards of study hospital, with the intent to evaluate all patients with respiratory failure for at least 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of deaths or hospital readmissions within three months of discharge | 3 months after hospital discharge
  Number of patients who died or were readmitted to the hospital within three month of hospital discharge

SECONDARY OUTCOMES:
Number of ER visits | 3 months after hospital discharge
  Number of visits to the emergency department within three months of hospital discharge.
Healthcare utilization | Within 3 months of hospital discharge
  Gather information about healthcare resources utilization. For example, readmission to hospital after discharge or visits with primary care doctor.
Cognitive Functional outcome as assessed by Montreal Cognitive Assessment (MoCA) - Blind Instrument | After 3 months of hospital discharge
  Using MoCA-Blind Instrument which assesses different types of cognitive abilities and can be administered via phone. Scores range from 0 to 22 points, with a score of 18 and higher generally considered normal.
Physical function outcome as assessed by Activity of Daily Living (ADL-Katz Index) | At 3 months after hospital discharge
  This will be assessed using the Activity of Daily Living (ADL-Katz Index) instrument. ADL evaluates functional status as a measurement of the patient's ability to perform activities of daily living. Each activity is rated as being completed independently or not. Scores range is 0-6 points, higher score is better.
Physical function outcome as assessed by Activity of Daily Living (ADL-Katz Index) | At 6 months after hospital discharge
  This will be assessed using the Activity of Daily Living (ADL-Katz Index) instrument. ADL evaluates functional status as a measurement of the patient's ability to perform activities of daily living. Each activity is rated as being completed independently or not. Scores range is 0-6 points, higher score is better.
Physical function outcome as assessed by Instrumental Activity of Daily Living (IADL-Lawton) | At 3 months after hospital discharge
  This will be assessed using the Instrumental Activity of Daily Living (IADL-Lawton) instrument. IADL evaluates independent living skills. Each activity has specific level of participation that can be selected. Scores range from 0 (low function, dependent) to 8 points (high function, independent).
Physical function outcome as assessed by Instrumental Activity of Daily Living (IADL-Lawton) | At 6 months after hospital discharge
  This will be assessed using the Instrumental Activity of Daily Living (IADL-Lawton) instrument. IADL evaluates independent living skills. Each activity has specific level of participation that can be selected. Scores range from 0 (low function, dependent) to 8 points (high function, independent).
Mental health Functional outcome as assessed by Hospital Anxiety and Depression Scale (HADS) | After 3 months of hospital discharge
  Using Hospital Anxiety and Depression Scale (HADS) instrument which scores for anxiety and depression, range: 0-21 points; lower score is better, with scores ≥8 points, indicating substantial symptoms.
Functional outcomes-Post Traumatic Stress Disorder (PTSD) | After 3 months of hospital discharge
  Using Impact of Event Scale-Revised (IES-R) instrument which is a 22-item self-report measure that assesses subjective distress caused by traumatic events. range: 0-4 points; lower score is better, with scores ≥1.6 indicating substantial symptoms. For this outcome mean or median scores can be reported along the with the proportion of patients above the threshold.
Coping or social support | After 3 months of hospital discharge
  Using Multidimensional Scale of Perceived Social Support (MSPSS) instrument which is a brief (12-item) tool designed to measure perceptions of support from three sources: Family, Friends, and a Significant Other. Each item is scored on a 7-point Likert scale (ranging from Very Strongly Disagree to Very Strongly Agree, with midpoint as Neutral). Higher scores indicate greater levels of social support.
Health related quality of life | At 3 months after hospital discharge
  Using EQ-5D instrument which is a standardized instrument for measuring generic health status. EQ-5D-5L consists a descriptive system and the EQ Visual Analogue scale (EQ VAS).
  The descriptive system comprises 5 dimensions; Mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each is rated with 5 levels of severity of problems: no problems, slight problems, moderate problems, severe problems, extreme problems. The visual analog scale ranges from 0 to 100 with higher scores reflecting better perceived current health-related quality of life state.
Health related quality of life | At 6 months after hospital discharge
  Using EQ-5D instrument which is a standardized instrument for measuring generic health status. EQ-5D-5L consists a descriptive system and the EQ Visual Analogue scale (EQ VAS).
  The descriptive system comprises 5 dimensions; Mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each is rated with 5 levels of severity of problems: no problems, slight problems, moderate problems, severe problems, extreme problems. The visual analog scale ranges from 0 to 100 with higher scores reflecting better perceived current health-related quality of life state.
Number of deaths within 6 Months after discharge | 6 months after hospital discharge
  Number of patients who died within six months of hospital discharge
Return to work | 6 month after hospital discharge
  Employment status within six month after hospital discharge. Including addition descriptions of return to work, for example, change in duties or change in effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel M Brown, MD, Principal Investigator — Intermountain Medical Center; James C Jackson, PsyD, Principal Investigator — Vanderbilt University
Locations (5):
- United States (5):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Vanderbilt University, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah
  - George Wahlen Salt Lake City Veterans Administration Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Undecided
Privacy Concerns

REFERENCES:
- [Derived] Bose S, Groat D, Stollings JL, Barney P, Dinglas VD, Goodspeed VM, Carmichael H, Mir-Kasimov M, Jackson JC, Needham DM, Brown SM, Sevin CM; APICS-01 Study Team. Prescription of potentially inappropriate medications after an intensive care unit stay for acute respiratory failure. Aust Crit Care. 2024 Nov;37(6):866-872. doi: 10.1016/j.aucc.2024.02.001. Epub 2024 Apr 29. PMID 38688808
- [Derived] Bose S, Groat D, Dinglas VD, Akhlaghi N, Banner-Goodspeed V, Beesley SJ, Greene T, Hopkins RO, Mir-Kasimov M, Sevin CM, Turnbull AE, Jackson JC, Needham DM, Brown SM; Addressing Post-Intensive Care Syndrome (APICS-01) Study Team. Association Between Unmet Nonmedication Needs After Hospital Discharge and Readmission or Death Among Acute Respiratory Failure Survivors: A Multicenter Prospective Cohort Study. Crit Care Med. 2023 Feb 1;51(2):212-221. doi: 10.1097/CCM.0000000000005709. Epub 2023 Jan 20. PMID 36661449
- [Derived] Akhlaghi N, Needham DM, Bose S, Banner-Goodspeed VM, Beesley SJ, Dinglas VD, Groat D, Greene T, Hopkins RO, Jackson J, Mir-Kasimov M, Sevin CM, Wilson E, Brown SM. Evaluating the association between unmet healthcare needs and subsequent clinical outcomes: protocol for the Addressing Post-Intensive Care Syndrome-01 (APICS-01) multicentre cohort study. BMJ Open. 2020 Oct 23;10(10):e040830. doi: 10.1136/bmjopen-2020-040830. PMID 33099499

DOCUMENTS (1):
  • Informed Consent Form (2019-07-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT03738774/ICF_000.pdf